CLINICAL TRIAL: NCT04464863
Title: Kinematic Analysis in Stroke Patients Using Microsoft Kinect and Akira Software: Kinect-Akira Movement Study
Acronym: KAM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Other Study IDs: KAM-Study (PI-3787)
Record Dates: First submitted 2020-06-11; First posted 2020-07-09 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-04

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Acute stroke patients during the first week of evolution
  Interventions: Other: Kinematic metrics
- Control: Age and sex 1:1 healthy participants
  Interventions: Other: Kinematic metrics

INTERVENTIONS:
Other: Kinematic metrics — kinematic metrics recorded with Kinect (register brand) and extracted with Akira (register brand)

SUMMARY:
In this prospective, unicentric, case-control study, the main aim is to analyze joint movement and walking patterns in patients with acute stroke with a marker-free motion capture system. Case group: Stroke patients who fulfill the inclusion criteria are invited to participate in the study during admission. The evaluation consists of a workout designed by expert rehabilitation physicians and neurologists that is performed by the patient in front of the Microsoft Kinect camera. The custom-built software Akira record the joint angles of body trunk and upper limbs during the workout. The kinematic data will be analyzed with a machine learning algorithm that classifies the participant according to the kinematic data in normal movement or impaired movement (with the degree of impairment) by age decade. Control group: healthy participants (without neurological or osteomuscular diseases) matched by age and sex with cases 1:1. The correlation between kinematic and clinical scales (NIHSS) and functional scales (modified Rankin Scale) will be analyzed. A secondary objective will be to analyze the predictive value of the kinematic measurements with the functional outcome at three months

ELIGIBILITY:
Inclusion Criteria:

* Acute Stroke patients (within the first week of index stroke)
* Neurological deficit present at the moment of the evaluation.
* Informed consent signed.

Exclusion Criteria:

* Clinical instability
* Aphasia or cognitive decline that prevents the understanding of the workout.
* Refuse to participate
* Previous neurological or osteomuscular conditions.
* Previous conditions with less than 3 months of expectancy of life.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Acute stroke patients and healthy controls, matched by age and sex. The inclusion and exclusion criteria are defined below
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2020-01-29 (Actual); Primary Completion 2021-01-29 (Estimated); Study Completion 2021-06-29 (Estimated)

PRIMARY OUTCOMES:
Kinematic metrics: join angles | The change between the first week of index stroke (acute phase) and at 3 months after index stroke
  The kinect camera together with the software Akira will be used to automatically measure the degree angle of the following body joints: shoulder in abduction, shoulder inflexion, elbow in extension and in flexion and the angle formed by the forearm and the trunk with the shoulder in abduction.
Kinematic metrics: movement acceleration | The change between the first week of index stroke (acute phase) and at 3 months after index stroke
  The kinect camera together with the software Akira will be used to automatically measure the acceleration of the following movements: shoulder abduction and shoulder flexion.
Kinematic metrics: movement pattern | The change between the first week of index stroke (acute phase) and at 3 months after index stroke
  The kinect camera together with the software Akira will be used to automatically measure the pattern of the following movements: trunk oscillation during standing position and during walking; and trunk oscillation during seating position with opened and closed eyes.

SECONDARY OUTCOMES:
Relationship of kinematic measures with the degree of disability after stroke. | At 3 months after the index stroke
  Correlation between the kinematic metrics described before (joint angles, movement acceleration and movement pattern) and the degree of disability, measured y the modified Rankin scale. The modified Rankin Scale (mRS) is a extensively use scale to measure dependency after stroke. The minimum value is 0 (no sequels or disability) and the maximum value is 6 (dead). The lower the score in the scale, the better is the outcome.

CONTACTS AND LOCATIONS:
Overall Officials: María Alonso de Leciñana, MD PhD, Study Director — Hospital Universitario La Paz, IdiPAZ
Locations (1):
- La Paz University Hospital, IdiPAZ, Madrid, Spain